CLINICAL TRIAL: NCT03659617
Title: Clinical, Radiographic and Histomorphotmetric Analysis of Healing Dynamics in Human Extraction Sockets Grafted With Bio-Oss Collagen®: A Prospective 3-year Post-loading Study
Brief Title: Healing Dynamics in Human Extraction Sockets Grafted With Bio-Oss Collagen®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Principal Investigator, Carlos Garaicoa Pazmino, Principal Investigator, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201806050
Record Dates: First submitted 2018-07-10; First posted 2018-09-06 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Tooth Loss
Keywords: alveolar bone; alveolar ridge; bone resorption; bone grafting; barrier membrane
MeSH Terms: conditions — Tooth Loss; Bone Resorption | interventions — Transplantation, Heterologous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors collecting the data and conducting the appropriate statistical analyses for all outcomes in the study will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Implant placement 3 mo. after tooth ext. (Experimental): Alveolar ridge preservation using xenograft (BioOss Collagen) and Implant placement 3 mo. after tooth ext.
  Interventions: Device: xenograft (BioOss Collagen)
- Implant placement 6 mo. after tooth ext. (Active Comparator): Alveolar ridge preservation using xenograft (BioOss Collagen) and Implant placement 6 mo. after tooth ext.
  Interventions: Device: xenograft (BioOss Collagen)
- Implant placement 9 mo. after tooth ext. (Active Comparator): Alveolar ridge preservation using xenograft (BioOss Collagen) and Implant placement 9 mo. after tooth ext.
  Interventions: Device: xenograft (BioOss Collagen)

INTERVENTIONS:
Device: xenograft (BioOss Collagen) — Alveolar ridge preservation using xenograft (BioOss Collagen) and implant placement at 3 different time intervals (3, 6 and 9 months)

SUMMARY:
The purpose of this study is to clinically, radiographically and histologically evaluate the healing sequence of post-extraction sockets grafted with Bio-Oss Collagen® at 3, 6 and 9 months following tooth extraction in single-rooted tooth sites.

Subjects with single rooted teeth planned for extraction and replacement with endosseous dental implants will be recruited for the study based on the eligibility criteria and will be divided in three groups (Groups 1, 2 and 3).A cone-beam computed tomography (CBCT) scan will be obtained and reviewed to prepare for the surgical approach and evaluate the ridge dimensions, the tooth planned for extraction as well as the adjacent sites. After tooth extraction, the socket will be grafted with Bio-Oss Collagen® and, depending on the morphology of the extraction sockets, a collagen matrix (Mucograft® seal) and/or a restorable collagen membrane (BioGide®)will be placed to cover and stabilize the graft. Patients will return at 2 and 6 weeks post-extraction to evaluate the healing. A second CBCT will be obtained 2 weeks prior to implant placement to evaluate the ridge dimensions and compare them to the baseline data. Implant placement will take place at 12, 24 and 36 after tooth extraction for Groups 1, 2 and 3 respectively. A bone core biopsy will be obtained at the time of implant placement and will be sent for histological analysis. Patients will return for a post-operative visit at two weeks. Clinical indices (probing depth, recession, bleeding upon probing, keratinized mucosa height, plaque and gingival index), patient reported outcomes and marginal bone levels via standardized periapical radiographs will be evaluated and recorded at baseline (no more than 30 days following delivery of final implant restoration) 1, 2 and 3 years post-loading.

DETAILED DESCRIPTION:
Patients participating in this study are expected to return to the University of Iowa College of Dentistry for a total of 12 visits. The estimated study length per subject will vary between 42 to 48 months depending on group allocation.

VISIT 1: Screening Subjects in need of extraction of a single-rooted tooth, except for lower incisors, that meet all the inclusion and none of the exclusion criteria will be eligible to participate. The purpose of the study, the duration and the potential risks and benefits will be explained in detailed to the patients. If the subject is interested in participating in the study, copies of the study outline and consent forms will be given to them. Medical and dental history form will be entered in patients' charts electronically, completed and signed by the subjects. Intra-oral scan will be obtained (multiple photos that comprise a 3-D impression)

VISIT 2: Tooth Extraction (TE) and Ridge Preservation via Socket Grafting Medical and dental histories will be reviewed and possible changes will be recorded. Intra-oral photographs of the sites of interest will be obtained. Clinical and radiographic examination of the sites involved in the study will be performed. A cone-beam computed tomography (CBCT) scan will be obtained and reviewed to prepare for the surgical approach and evaluate the tooth planned for extraction as well as the adjacent sites for pathology and neighboring sensitive anatomic structures that can alter the proposed treatment plan. Digital intra-oral scanning of the area of interest will be performed using the Planmeca Emerald (TM) scanner. The subject will sign the surgical consent form. After administration of local anesthesia, the tooth will be extracted as less traumatically as possible, without flap reflection. Following tooth extraction, the socket walls will be clinically evaluated for the existence of dehiscences or fenestrations. Sites presenting a bony defect affecting >50% of the total wall height will be excluded. Sockets will be grafted with Bio-Oss Collagen®, BioGide® will be utilized if indicated for the treatment for a dehiscence and the coronal part will be covered with a collagen matrix (Mucograft Seal®). Stabilizing sutures will be applied to maintain the collagen matrix adequately in place. Written and verbal post-operative instructions will be given to the patients. They will be instructed to avoid any mechanical disturbance in the area for two weeks. Patients will be asked to use a mouthwash containing 0.12% of chlorhexidine gluconate twice a day, thirty seconds at a time, avoiding any eating or drinking for 30 minutes after rinsing, starting 48 hours after the baseline intervention. Post-operative medication (antibiotics, analgesics, NSAIDs) will be prescribed on an individual basis.

VISIT 3 (TE + 1 week) & VISIT 4 (TE + 2 weeks): Postops Medical and dental histories will be reviewed and possible changes will be recorded. Intra-oral photographs and Intra-oral scan (multiple photos that comprise a 3-D impression) of the sites of interest will be obtained. Visual assessment of the healing status will be made using a WHI. Patients will be asked to report their pain using a Visual Analog Scale (VAS). Sutures will be removed at either of the two visits. Sites will be debrided, if necessary. and oral hygiene instructions will be reviewed.

VISIT 5: Post-op (TE + 6 weeks) Medical and dental histories will be reviewed and possible changes will be recorded. Intra-oral photographs and Intra-oral scan will be obtained (multiple photos that comprise a 3-D impression) of the sites of interest will be obtained. Visual assessment of the healing status will be made using a WHI. Patients will be asked to report their pain using a VAS. Gentle plaque debridement will be provided and oral hygiene instructions will be reviewed.

VISIT 6: Follow-up and second CBCT scan Group 1 (TE + 10 weeks) Group 2 (TE + 22 weeks) Group 3 (TE + 34 weeks) Medical and dental histories will be reviewed and updated, if necessary. Intra-oral pictures of the surgical sites will be obtained. At this visit, a second segmental CBCT scan will be obtained for all patients, using the same settings employed at baseline. Images will be used to analyze and compare the ridge dimensions to those obtained at baseline as well as in terms of adequacy for dental implant placement. Intra-oral scan will be obtained (multiple photos that comprise a 3-D impression).

VISIT 7: Implant Placement and Bone Core Biopsy Harvesting Group 1 (TE + 12 weeks) Group 2 (TE + 24 weeks) Group 3 (TE + 36 weeks) Medical and dental histories will be reviewed and possible changes will be recorded. Intra-oral photographs of the sites of interest will be obtained. Digital intra-oral scanning of the area of interest will be performed using the Planmeca Emerald (TM) scanner. Implant placement will be done per standard procedure. A trephine drill of 2.5 mm diameter, or wider, will be used to harvest a bone core for histologic and µ-CT analyses. The bone core will be immediately submerged in a solution of 10% neutral buffered formalin (NBF). The selection of the implant system and dimensions will depend on the surgical and restorative needs of each individual case. Osteotomies and implant placement will be done following the manufacturer's recommendations. A final periapical radiograph will be obtained to verify correct implant position and angulation. Depending on the buccal bone and soft tissue thickness, ancillary soft tissue augmentation, bone augmentation or a combination of both may be indicated. If adequate primary stability is achieved and a one-stage approach is feasible, a healing abutment will be placed. If a two-stage procedure is indicated, a cover screw will be placed and the implant will be submerged. At the end of the appointment, written and verbal post-operative instructions will be given to the patients.

VISIT 8: Post-op (Implant Placement + 2 weeks) Medical and dental histories will be reviewed and possible changes will be recorded. Intra-oral photographs of the sites of interest will be obtained. Sutures will be removed. Visual assessment of the healing status will be made using a WHI. Patients will be asked to report their pain using a VAS. The sites will be debrided and oral hygiene instructions will be reviewed. Upon completion of this visit, the patient will be referred to the restorative dentist to complete the restorative part of the treatment.

VISIT 9: Baseline Implant Follow-up (No more than 30 days after delivery of final restoration) Medical and dental histories will be reviewed and possible changes will be recorded. Intra-oral photographs of the sites of interest will be obtained. Digital intra-oral scanning of the area of interest will be performed using the Planmeca Emerald (TM) scanner. Patients will be asked to report their level of satisfaction in terms of function, comfort and esthetics (PROMs). The sites will be inspected, deplaqued, if necessary, and oral hygiene instructions will be reviewed. Clinical parameters will be recorded (i.e. probing depth, recession respective to the incisal/occlusal plane, bleeding upon probing, keratinized mucosa height, plaque and gingival index). A standardized periapical radiograph will be obtained to assess marginal bone levels.

VISIT 10: Implant Follow-up #1 (1 year after delivery of final restoration) Medical and dental histories will be reviewed and possible changes will be recorded. Intra-oral photographs of the sites of interest will be obtained. Digital intra-oral scanning of the area of interest will be performed using the Planmeca Emerald (TM) scanner. Patients will be asked to report their level of satisfaction in terms of function, comfort and esthetics (PROMs). The sites will be inspected, de-plaqued, if necessary, and oral hygiene instructions will be reviewed. Clinical parameters will be recorded (i.e. probing depth, recession respective to the incisal/occlusal plane, bleeding upon probing, keratinized mucosa height, plaque and gingival index). A standardized periapical radiograph will be obtained to assess marginal bone levels.

VISIT 11: Implant Follow-up #2 (2 years after delivery of final restoration) Medical and dental histories will be reviewed and possible changes will be recorded. Intra-oral photographs of the sites of interest will be obtained. Digital intra-oral scanning of the area of interest will be performed using the Planmeca Emerald (TM) scanner. Patients will be asked to report their level of satisfaction in terms of function, comfort and esthetics (PROMs). The sites will be inspected, de-plaqued, if necessary, and oral hygiene instructions will be reviewed. Clinical parameters will be recorded (i.e. probing depth, recession respective to the incisal/occlusal plane, bleeding upon probing, keratinized mucosa height, plaque and gingival index). A standardized periapical radiograph will be obtained to assess marginal bone levels.

VISIT 12: Implant Follow-up #3 (3 years after delivery of final restoration) Medical and dental histories will be reviewed and possible changes will be recorded. Intra-oral photographs of the sites of interest will be obtained. Digital intra-oral scanning of the area of interest will be performed using the Planmeca Emerald (TM) scanner. Patients will be asked to report their level of satisfaction in terms of function, comfort and esthetics (PROMs). The sites will be inspected, de-plaqued, if necessary, and oral hygiene instructions will be reviewed. Clinical parameters will be recorded (i.e. probing depth, recession respective to the incisal/occlusal plane, bleeding upon probing, keratinized mucosa height, plaque and gingival index). A standardized periapical radiograph will be obtained to assess marginal bone levels.

This is planned to be the final study visit.

ELIGIBILITY:
Inclusion Criteria:

* May be either male or female
* Age: 18 years or older
* Subjects with a single-rooted tooth (except mandibular incisors) indicated for extraction
* Extractions socket walls should either be intact or have no more than one bony wall (buccal or lingual) dehiscence extending no more than 50% of the total bony wall height
* Must be in adequate physical and mental health to undergo routine dental treatment including the surgical procedures associated tooth extraction and implant placement
* Subjects' treatment plan must include replacement of the tooth to be extracted with dental implant supported fixed restoration
* Subjects must have read, understood and signed an informed consent form

Exclusion Criteria:

* Mandibular incisors
* Acute infection associated with the tooth to be extracted or with adjacent teeth
* History of significant heart, stomach, liver, kidney, blood, immune system disease, or other organ impairment or systemic diseases that would prevent undergoing the proposed treatment or may result in compromised healing (e.g. poorly controlled diabetes, active heavy tobacco use [>10 cigs/day])
* Subjects with uncontrolled and/or severe metabolic bone diseases or disorders, such as osteoporosis, thyroid disorders or Paget's disease
* Subjects taking any medication or supplement known to largely influence bone metabolism, such as IV bisphosphonates, long-term history of oral bisphosphonates or chronic intake of glucocorticoids
* Pregnant women or nursing mothers
* Subjects that are unwilling or unable to sign the informed consent
* History of lack of compliance with dental visits
* Subjects unwilling to return for the required number of visits

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Implant survival | 3 years post implant loading
  did the implant survive

SECONDARY OUTCOMES:
% of vital bone via histomorphotmetric evaluation of bone core biopsies at 3 months | 3 months
  % of vital bone
% of vital bone via histomorphotmetric evaluation of bone core biopsies at 6 months | 6 months
  % of vital bone
% of vital bone via histomorphotmetric evaluation of bone core biopsies at 9 months | 9 months
  % of vital bone
Amount of mineralization via micro-CT analysis 3 months | 3 months
  Amount of mineralization
Amount of mineralization via micro-CT analysis 6 months | 6 months
  Amount of mineralization
Amount of mineralization via micro-CT analysis 9 months | 9 months
  Amount of mineralization
Linear Dimensional alterations of the alveolar ridge from the time of tooth extraction to the time of implant placement (3 months) | 3 months
  Clinical and radiographic (via CBCT) assessment. The buccal - lingual ridge width at the time of the extraction will be measured clinically using a periodontal probe (UNC-15) and prior to implant placement (3-months). The same measurements will be performed radiographically through the CBCTs taken prior to tooth extraction and prior to implant placement, utilizing a CBCT viewer software. The linear vertical alterations will be used utilizing the same methods, using fiduciary anatomical landmarks. Superimposition of the digital files obtained from the intra-oral scanner will be utilized to verify these changes clinically.
Linear dimensional alterations of the alveolar ridge from the time of tooth extraction to the time of implant placement (6 months) | 6 months
  Clinical and radiographic (via CBCT) assessment. The buccal - lingual ridge width at the time of the extraction will be measured clinically using a periodontal probe (UNC-15) and prior to implant placement (6-months). The same measurements will be performed radiographically through the CBCTs taken prior to tooth extraction and prior to implant placement, utilizing a CBCT viewer software. The linear vertical alterations will be used utilizing the same methods, using fiduciary anatomical landmarks. Superimposition of the digital files obtained from the intra-oral scanner will be utilized to verify these changes clinically.
Linear dimensional alterations of the alveolar ridge from the time of tooth extraction to the time of implant placement (9 months) | 9 months
  Clinical and radiographic (via CBCT) assessment. The buccal - lingual ridge width at the time of the extraction will be measured clinically using a periodontal probe (UNC-15) and prior to implant placement (9-months). The same measurements will be performed radiographically through the CBCTs taken prior to tooth extraction and prior to implant placement, utilizing a CBCT viewer software. The linear vertical alterations will be used utilizing the same methods, using fiduciary anatomical landmarks. Superimposition of the digital files obtained from the intra-oral scanner will be utilized to verify these changes clinically.
Assessment of the mucosal maturation of the extraction sites after the use of Mucograft Seal® @ 1 week, using a wound healing index (1-3 scale rating) | 1 week following tooth extraction and alveolar ridge preservation
  Wound Healing Index. 1-3 scale rating: 1) Uneventful Healing, 2) Normal healing with moderate soft tissue inflammation, erythema but no suppuration and 3) poor wound healing with significant signs of clinical inflammation and/or suppuration
Assessment of the mucosal maturation of the extraction sites after the use of Mucograft Seal® @ 2 weeks, using a wound healing index (1-3 scale rating) | 2 weeks following tooth extraction and alveolar ridge preservation
  Wound Healing Index.1-3 scale rating: 1) Uneventful Healing, 2) Normal healing with moderate soft tissue inflammation, erythema but no suppuration and 3) poor wound healing with significant signs of clinical inflammation and/or suppuration
Assessment of the mucosal maturation of the extraction sites after the use of Mucograft Seal® @ 6 weeks, using a wound healing index (1-3 scale rating) | 6 weeks following tooth extraction and alveolar ridge preservation
  Wound Healing Index. 1-3 scale rating: 1) Uneventful Healing, 2) Normal healing with moderate soft tissue inflammation, erythema but no suppuration and 3) poor wound healing with significant signs of clinical inflammation and/or suppuration
Assessment of the mucosal maturation following implant placement, using a wound healing index (1-3 scale rating) | 2 weeks following dental implant placement
  Wound Healing Index. 1-3 scale rating: 1) Uneventful Healing, 2) Normal healing with moderate soft tissue inflammation, erythema but no suppuration and 3) poor wound healing with significant signs of clinical inflammation and/or suppuration
Patient reported outcomes (pain) 1 week following tooth extraction, using a Visual Analog Score for pain (0-100) | 1 week following tooth extraction and alveolar ridge preservation
  Visual Analog Score for pain (0-100, with 0 representing no pain, and 100 very severe pain, described as "worse pain imaginable").
Patient reported outcomes (pain) 2 weeks following tooth extraction, using a Visual Analog Score for pain (0-100) | 2 weeks following tooth extraction and alveolar ridge preservation
  Visual Analog Score for pain (0-100, with 0 representing no pain, and 100 very severe pain, described as "worse pain imaginable").
Patient reported outcomes (pain) 6 weeks following tooth extraction, using a Visual Analog Score for pain (0-100) | 6 weeks following tooth extraction and alveolar ridge preservation
  Visual Analog Score for pain (0-100, with 0 representing no pain, and 100 very severe pain, described as "worse pain imaginable").
Patient reported outcomes (pain) 2 weeks following implant placement, using a Visual Analog Score for pain (0-100) | 2 weeks following implant placement
  Visual Analog Score for pain (0-100, with 0 representing no pain, and 100 very severe pain, described as "worse pain imaginable").
Patient reported outcomes (patient satisfaction), using a Visual Analog Scale (0-100) | Up to 30 days post implant crown delivery
  The patients will be asked to rate their satisfaction in terms of function, comfort and esthetics, using a Visual Analog Scale (0-100, with 0 meaning "not at satisfied at all" and 100 corresponding to "perfectly satisfied").
Marginal bone level changes | 3 years post implant crown delivery
  measured in mm based on standardized intro-oral radiographs

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Garaicoa Pazmino, DDS, Principal Investigator — University of Iowa
Locations (1):
- The University of Iowa College of Dentistry and Dental Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrams L. Augmentation of the deformed residual edentulous ridge for fixed prosthesis. Compend Contin Educ Gen Dent. 1980 May-Jun;1(3):205-13. No abstract available. PMID 6950834
- [Background] Aghaloo TL, Misch C, Lin GH, Iacono VJ, Wang HL. Bone Augmentation of the Edentulous Maxilla for Implant Placement: A Systematic Review. Int J Oral Maxillofac Implants. 2016;31 Suppl:s19-30. doi: 10.11607/jomi.16suppl.g1. PMID 27228250
- [Background] Aghaloo TL, Moy PK. Which hard tissue augmentation techniques are the most successful in furnishing bony support for implant placement? Int J Oral Maxillofac Implants. 2007;22 Suppl:49-70. PMID 18437791
- [Background] Alkan EA, Parlar A, Yildirim B, Senguven B. Histological comparison of healing following tooth extraction with ridge preservation using enamel matrix derivatives versus Bio-Oss Collagen: a pilot study. Int J Oral Maxillofac Surg. 2013 Dec;42(12):1522-8. doi: 10.1016/j.ijom.2013.06.002. Epub 2013 Jul 8. PMID 23845297
- [Background] Amler MH. The time sequence of tissue regeneration in human extraction wounds. Oral Surg Oral Med Oral Pathol. 1969 Mar;27(3):309-18. doi: 10.1016/0030-4220(69)90357-0. No abstract available. PMID 5251474
- [Background] Araujo M, Linder E, Wennstrom J, Lindhe J. The influence of Bio-Oss Collagen on healing of an extraction socket: an experimental study in the dog. Int J Periodontics Restorative Dent. 2008 Apr;28(2):123-35. PMID 18546808
- [Background] Araujo MG, da Silva JCC, de Mendonca AF, Lindhe J. Ridge alterations following grafting of fresh extraction sockets in man. A randomized clinical trial. Clin Oral Implants Res. 2015 Apr;26(4):407-412. doi: 10.1111/clr.12366. Epub 2014 Mar 12. PMID 24621203
- [Background] Araujo MG, Liljenberg B, Lindhe J. Dynamics of Bio-Oss Collagen incorporation in fresh extraction wounds: an experimental study in the dog. Clin Oral Implants Res. 2010 Jan;21(1):55-64. doi: 10.1111/j.1600-0501.2009.01854.x. PMID 20070748
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] Avila-Ortiz G, Elangovan S, Kramer KW, Blanchette D, Dawson DV. Effect of alveolar ridge preservation after tooth extraction: a systematic review and meta-analysis. J Dent Res. 2014 Oct;93(10):950-8. doi: 10.1177/0022034514541127. Epub 2014 Jun 25. PMID 24966231
- [Background] Barone A, Aldini NN, Fini M, Giardino R, Calvo Guirado JL, Covani U. Xenograft versus extraction alone for ridge preservation after tooth removal: a clinical and histomorphometric study. J Periodontol. 2008 Aug;79(8):1370-7. doi: 10.1902/jop.2008.070628. PMID 18672985
- [Background] Beitlitum I, Artzi Z, Nemcovsky CE. Clinical evaluation of particulate allogeneic with and without autogenous bone grafts and resorbable collagen membranes for bone augmentation of atrophic alveolar ridges. Clin Oral Implants Res. 2010 Nov;21(11):1242-50. doi: 10.1111/j.1600-0501.2010.01936.x. PMID 20572833
- [Background] Boyne PJ. Osseous repair of the postextraction alveolus in man. Oral Surg Oral Med Oral Pathol. 1966 Jun;21(6):805-13. doi: 10.1016/0030-4220(66)90104-6. No abstract available. PMID 5219671
- [Background] Canullo L, Iurlaro G, Iannello G. Double-blind randomized controlled trial study on post-extraction immediately restored implants using the switching platform concept: soft tissue response. Preliminary report. Clin Oral Implants Res. 2009 Apr;20(4):414-20. doi: 10.1111/j.1600-0501.2008.01660.x. PMID 19298296
- [Background] Cardaropoli D, Tamagnone L, Roffredo A, Gaveglio L. Evaluation of Dental Implants Placed in Preserved and Nonpreserved Postextraction Ridges: A 12-Month Postloading Study. Int J Periodontics Restorative Dent. 2015 Sep-Oct;35(5):677-85. doi: 10.11607/prd.2309. PMID 26357697
- [Background] Chappuis V, Engel O, Shahim K, Reyes M, Katsaros C, Buser D. Soft Tissue Alterations in Esthetic Postextraction Sites: A 3-Dimensional Analysis. J Dent Res. 2015 Sep;94(9 Suppl):187S-93S. doi: 10.1177/0022034515592869. Epub 2015 Jun 30. PMID 26130259
- [Background] Danan M, Degrange M, Vaideanu T, Brion M. Immediate replacement of a maxillary central incisor associated with severe facial bone loss: use of Bio-Oss collagen--case report. Int J Periodontics Restorative Dent. 2003 Oct;23(5):491-7. PMID 14620123
- [Background] Degidi M, Daprile G, Nardi D, Piattelli A. Buccal bone plate in immediately placed and restored implant with Bio-Oss((R)) collagen graft: a 1-year follow-up study. Clin Oral Implants Res. 2013 Nov;24(11):1201-5. doi: 10.1111/j.1600-0501.2012.02561.x. Epub 2012 Aug 13. PMID 22882574
- [Background] Discepoli N, Vignoletti F, Laino L, de Sanctis M, Munoz F, Sanz M. Fresh extraction socket: spontaneous healing vs. immediate implant placement. Clin Oral Implants Res. 2015 Nov;26(11):1250-5. doi: 10.1111/clr.12447. Epub 2014 Jul 17. PMID 25041072
- [Background] Evian CI, Rosenberg ES, Coslet JG, Corn H. The osteogenic activity of bone removed from healing extraction sockets in humans. J Periodontol. 1982 Feb;53(2):81-5. doi: 10.1902/jop.1982.53.2.81. PMID 6950085
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Fu JH, Wang HL. Horizontal bone augmentation: the decision tree. Int J Periodontics Restorative Dent. 2011 Jul-Aug;31(4):429-36. PMID 21837309
- [Background] Heberer S, Al-Chawaf B, Hildebrand D, Nelson JJ, Nelson K. Histomorphometric analysis of extraction sockets augmented with Bio-Oss Collagen after a 6-week healing period: a prospective study. Clin Oral Implants Res. 2008 Dec;19(12):1219-25. doi: 10.1111/j.1600-0501.2008.01617.x. No abstract available. PMID 19040436
- [Background] Heinemann F, Hasan I, Schwahn C, Bourauel C, Mundt T. Bone level change of extraction sockets with Bio-Oss collagen and implant placement: a clinical study. Ann Anat. 2012 Nov;194(6):508-12. doi: 10.1016/j.aanat.2011.11.012. Epub 2011 Dec 23. PMID 22244384
- [Background] Iasella JM, Greenwell H, Miller RL, Hill M, Drisko C, Bohra AA, Scheetz JP. Ridge preservation with freeze-dried bone allograft and a collagen membrane compared to extraction alone for implant site development: a clinical and histologic study in humans. J Periodontol. 2003 Jul;74(7):990-9. doi: 10.1902/jop.2003.74.7.990. PMID 12931761
- [Background] Jung RE, Philipp A, Annen BM, Signorelli L, Thoma DS, Hammerle CH, Attin T, Schmidlin P. Radiographic evaluation of different techniques for ridge preservation after tooth extraction: a randomized controlled clinical trial. J Clin Periodontol. 2013 Jan;40(1):90-8. doi: 10.1111/jcpe.12027. Epub 2012 Nov 19. PMID 23163915
- [Background] Kao RT. Strategic extraction: a paradigm shift that is changing our profession. J Periodontol. 2008 Jun;79(6):971-7. doi: 10.1902/jop.2008.070551. PMID 18533770
- [Background] Kuchler U, von Arx T. Horizontal ridge augmentation in conjunction with or prior to implant placement in the anterior maxilla: a systematic review. Int J Oral Maxillofac Implants. 2014;29 Suppl:14-24. doi: 10.11607/jomi.2014suppl.g1.1. PMID 24660187
- [Background] Lekovic V, Kenney EB, Weinlaender M, Han T, Klokkevold P, Nedic M, Orsini M. A bone regenerative approach to alveolar ridge maintenance following tooth extraction. Report of 10 cases. J Periodontol. 1997 Jun;68(6):563-70. doi: 10.1902/jop.1997.68.6.563. PMID 9203100
- [Background] Meloni SM, Tallarico M, Lolli FM, Deledda A, Pisano M, Jovanovic SA. Postextraction socket preservation using epithelial connective tissue graft vs porcine collagen matrix. 1-year results of a randomised controlled trial. Eur J Oral Implantol. 2015 Spring;8(1):39-48. PMID 25738178
- [Background] Nart J, Barallat L, Jimenez D, Mestres J, Gomez A, Carrasco MA, Violant D, Ruiz-Magaz V. Radiographic and histological evaluation of deproteinized bovine bone mineral vs. deproteinized bovine bone mineral with 10% collagen in ridge preservation. A randomized controlled clinical trial. Clin Oral Implants Res. 2017 Jul;28(7):840-848. doi: 10.1111/clr.12889. Epub 2016 Jun 22. PMID 27335267
- [Background] Nemcovsky CE, Serfaty V. Alveolar ridge preservation following extraction of maxillary anterior teeth. Report on 23 consecutive cases. J Periodontol. 1996 Apr;67(4):390-5. doi: 10.1902/jop.1996.67.4.390. PMID 8708965
- [Background] Nevins M, Camelo M, De Paoli S, Friedland B, Schenk RK, Parma-Benfenati S, Simion M, Tinti C, Wagenberg B. A study of the fate of the buccal wall of extraction sockets of teeth with prominent roots. Int J Periodontics Restorative Dent. 2006 Feb;26(1):19-29. PMID 16515093
- [Background] Nevins ML, Camelo M, Lynch SE, Schenk RK, Nevins M. Evaluation of periodontal regeneration following grafting intrabony defects with bio-oss collagen: a human histologic report. Int J Periodontics Restorative Dent. 2003 Feb;23(1):9-17. PMID 12617364
- [Background] Nevins ML, Camelo M, Rebaudi A, Lynch SE, Nevins M. Three-dimensional micro-computed tomographic evaluation of periodontal regeneration: a human report of intrabony defects treated with Bio-Oss collagen. Int J Periodontics Restorative Dent. 2005 Aug;25(4):365-73. PMID 16089044
- [Background] Orth CF. A modification of the connective tissue graft procedure for the treatment of type II and type III ridge deformities. Int J Periodontics Restorative Dent. 1996 Jun;16(3):266-77. PMID 9084312
- [Background] Reddy KP, Nayak DG, Uppoor AS. A clinical evaluation of anorganic bovine bone graft plus 10% collagen with or without a barrier in the treatment of class II furcation defects. J Contemp Dent Pract. 2006 Feb 15;7(1):60-70. PMID 16491148
- [Background] Roccuzzo M, Gaudioso L, Bunino M, Dalmasso P. Long-term stability of soft tissues following alveolar ridge preservation: 10-year results of a prospective study around nonsubmerged implants. Int J Periodontics Restorative Dent. 2014 Nov-Dec;34(6):795-804. doi: 10.11607/prd.2133. PMID 25411735
- [Background] Roccuzzo M, Gaudioso L, Lungo M, Dalmasso P. Surgical therapy of single peri-implantitis intrabony defects, by means of deproteinized bovine bone mineral with 10% collagen. J Clin Periodontol. 2016 Mar;43(3):311-8. doi: 10.1111/jcpe.12516. Epub 2016 Mar 9. PMID 26800389
- [Background] Saadoun AP. Periodontal and restorative considerations in strategic extractions. Compend Contin Educ Dent (Lawrenceville). 1981 Jan-Feb;2(1):48-55. No abstract available. PMID 6950850
- [Background] Scheyer ET, Heard R, Janakievski J, Mandelaris G, Nevins ML, Pickering SR, Richardson CR, Pope B, Toback G, Velasquez D, Nagursky H. A randomized, controlled, multicentre clinical trial of post-extraction alveolar ridge preservation. J Clin Periodontol. 2016 Dec;43(12):1188-1199. doi: 10.1111/jcpe.12623. Epub 2016 Oct 21. PMID 27617409
- [Background] Schropp L, Wenzel A, Kostopoulos L, Karring T. Bone healing and soft tissue contour changes following single-tooth extraction: a clinical and radiographic 12-month prospective study. Int J Periodontics Restorative Dent. 2003 Aug;23(4):313-23. PMID 12956475
- [Background] Seibert JS, Louis JV. Soft tissue ridge augmentation utilizing a combination onlay-interpositional graft procedure: a case report. Int J Periodontics Restorative Dent. 1996 Aug;16(4):310-21. PMID 9242099
- [Background] Tonetti MS, Steffen P, Muller-Campanile V, Suvan J, Lang NP. Initial extractions and tooth loss during supportive care in a periodontal population seeking comprehensive care. J Clin Periodontol. 2000 Nov;27(11):824-31. doi: 10.1034/j.1600-051x.2000.027011824.x. PMID 11073325
- [Background] Trevisiol L, Nocini PF, Albanese M, Sbarbati A, D'Agostino A. Grafting of large mandibular advancement with a collagen-coated bovine bone (Bio-Oss Collagen) in orthognathic surgery. J Craniofac Surg. 2012 Sep;23(5):1343-8. doi: 10.1097/SCS.0b013e3182646c3a. PMID 22948619
- [Derived] Couso-Queiruga E, Weber HA, Garaicoa-Pazmino C, Barwacz C, Kalleme M, Galindo-Moreno P, Avila-Ortiz G. Influence of healing time on the outcomes of alveolar ridge preservation using a collagenated bovine bone xenograft: A randomized clinical trial. J Clin Periodontol. 2023 Feb;50(2):132-146. doi: 10.1111/jcpe.13744. Epub 2022 Nov 18. PMID 36345818